CLINICAL TRIAL: NCT06364124
Title: Effects of PCSK-9 Inhibitor Treatment Prior to Undergoing Primary Percutaneous Coronary Intervention in Patients With ST-segment Elevation Myocardial Infarction: A Single-center，Randomized,Open-label Trial
Brief Title: Effects of PCSK-9 Inhibitor Treatment Prior to Undergoing Primary Percutaneous Coronary Intervention in Patients With ST-segment Elevation Myocardial Infarction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Luhe Hospital (Other)
Responsible Party: Principal Investigator, Jincheng Guo, Clinical Professor, Beijing Luhe Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MR-11-23-035852
Record Dates: First submitted 2024-04-01; First posted 2024-04-15 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: STEMI
Keywords: evolocumab; STEMI; LDL-C
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm: standard post-treatment for STEMI and Evolocumab (Experimental): The intervention group will receive a preoperative subcutaneous injection of Evolocumab (420mg) and standard post-treatment for STEMI
  Interventions: Drug: evolocumab; Procedure: standard post-treatment for STEMI
- Control arm: standard post-treatment for STEMI (Active Comparator): Standard post-treatment for STEMI
  Interventions: Procedure: standard post-treatment for STEMI

INTERVENTIONS:
Drug: evolocumab — Preoperative subcutaneous injection of Evolocumab (420mg)，Atorvastatin 40mg per day
  Other Names: repatha
  Arms: Treatment arm: standard post-treatment for STEMI and Evolocumab
Procedure: standard post-treatment for STEMI — standard post-treatment for STEMI

SUMMARY:
Acute ST-segment elevation myocardial infarction (STEMI) is a common manifestation of cardiovascular emergencies. Percutaneous coronary intervention (PCI) and guideline-recommended pharmacotherapy have reduced mortality rates associated with STEMI, but the incidence of recurrent ischemic events, particularly early ischemic events, remains high. Current research suggests that low-density lipoprotein cholesterol (LDL-C) levels not meeting guideline-recommended levels and inflammation are closely related to early recurrent ischemic events. Evolocumab, a proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitor, rapidly and effectively reduces LDL-C levels and suppresses inflammation. Long-term use in patients with acute coronary syndromes can reverse atherosclerosis and improve prognosis. However, data on its use in STEMI patients are limited, particularly regarding the cardioprotective effects of preoperative administration of 420mg evolocumab subcutaneous injection. This study aims to evaluate the effects of administering evolocumab 420mg before emergency PCI on lipid profiles, inflammatory markers, myocardial injury, and short-term prognosis in STEMI patients through a single-center, randomized, open-label study. It aims to provide theoretical evidence for further reducing the risk of recurrent cardiovascular events in STEMI and identifying more optimized treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* All patients are selected from the Cardiology Department of Beijing Luhe Hospital and have undergone direct PCI treatment for STEMI.
* STEMI patients must meet the following criteria:

  1. Chest pain duration ≥ 30 minutes, with ST-segment elevation ≥ 0.1 mV in adjacent two leads on the electrocardiogram.
  2. Onset within 24 hours.
  3. Aged between 18 and 80 years.
  4. Signed informed consent form.

Exclusion Criteria:

* Hemodynamically unstable or Killip grade ≥ 2.
* Severe renal insufficiency: Glomerular filtration rate < 30 ml/min/1.73m^2.
* Active liver disease or liver dysfunction: AST or ALT levels > 3 times the upper limit of normal.
* Known allergy to any drug used in the study.
* Previous or planned use of PCSK9 inhibitors.
* Suspected stress cardiomyopathy or acute pericarditis.
* Malignant tumors requiring treatment or other severe systemic diseases.
* Pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Average percent change from baseline in LDL-C levels to discharge and day 30 | 30 days

SECONDARY OUTCOMES:
Average percent change from baseline in total cholesterol, high-density lipoprotein cholesterol, triglycerides, apolipoprotein A and apolipoprotein B to discharge and day 30 | 30 days
Average percent change from baseline in MMP-9, CSF-1, IL-18R1 to discharge and day 30 | 30 days
Number of cardiovascular events to day 30 | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing luhe hospital, Beijing, China